CLINICAL TRIAL: NCT05615155
Title: Efficacy of C-PRF Versus i-PRF on Gingival Thickness & Keratinized Tissue Width in Subjects With Thin Gingival Biotype: ( Split Mouth Controlled Clinical Trials)
Brief Title: Efficacy of C-PRF vs i-PRF in Thin Gingival Biotype Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sajjad Ahmed Shakir (Other)
Responsible Party: Sponsor-Investigator, Sajjad Ahmed Shakir, bachelor of dental surgery, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Sajjad Ahmed Shakir
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Thin Gingival Biotype
MeSH Terms: interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- i-PRF (Experimental): The sides of the mouth that will be injected with injectable-Platelets Rich Fibrin
  Interventions: Other: Platelets Rich Fibrin (i-PRF / C-PRF)
- C-PRF (Experimental): The sides of the mouth that will be injected with Concentrated-Platelets Rich Fibrin
  Interventions: Other: Platelets Rich Fibrin (i-PRF / C-PRF)

INTERVENTIONS:
Other: Platelets Rich Fibrin (i-PRF / C-PRF) — one site of the mouth will be injected with i-PRF and the other site will be injected with C-PRF

SUMMARY:
Randomized split mouth clinical trials study focused on comparing the efficacy of i-prf versus c-prf injections on gingival thickness and keratinized tissue width in subjects with thin gingival biotype.

DETAILED DESCRIPTION:
Randomized split mouth clinical trials study focused on comparing the efficacy of i-prf versus c-prf injections on gingival thickness and keratinized tissue width in subjects with thin gingival biotype.

Gingival biotype is an important clinical parameter that plays an important role in determining the gingival health in the future and the possibility of developing gingival recession or other gingival unhealthy condition that is related to thin gingival biotype.

Gingival biotype is consist of gingival thickness and keratinized tissue width, and its either thin or thick, and the later is more favourable to withstand the developing of gingival diseases and unhealthy condition, with this study we compare the effect of i-PRF injection which is approved in many previous clinical trials that it affects the gingival biotype and increases gingival thickness and the keratinized tissue width, and compare it to newly developed PRF generation (C-PRF) which is Concentrated Platelet Rich Fibrin.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and no systemic disease or pregnancy.
2. Non-smoker.
3. Subjects with clinically healthy intact periodontium; bleeding on probing (BOP)<10%, probing pocket depth (PPD)≤3mm, intact periodontium (no probing attachment loss). (Chapple et al., 2018).
4. Four non-adjacent sites of anterior region with thin gingival biotype (GT ≤ 1mm). (Patrick H. et al., 2018).
5. No malocclusion, crowding, filling, missing or supernumerary mandibular anterior teeth.
6. No blood-borne conditions.
7. Any symptoms of recent acute illness e.g., COVID-19.

Exclusion Criteria

1. Active orthodontic treatment.
2. Previous periodontal surgery.
3. Use of blood thinners.
4. Use of any drugs that might lead to gingival enlargement.
5. Attrition.
6. Gingival Recession.
7. Thick gingival biotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
measure the mean differences gain of GT&KTW | baseline and 3 months
  the increase in gingival thickness and keratinized tissue width after the injection of prf concentrates.

SECONDARY OUTCOMES:
measure the mean difference gain of GT&KTW | baseline and 1 month
  the increase in gingival thickness and keratinized tissue width after the injection of prf concentrates.

CONTACTS AND LOCATIONS:
Overall Officials: Sajjad ah Shakir, BDS, Principal Investigator — University of Baghdad
Locations (1):
- University of Baghdad, Baghdad, Alresafa, Iraq

IPD SHARING:
Plan to Share IPD: No
the study will be published and shared for other researchers in medical journals.

DOCUMENTS (1):
  • Study Protocol (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT05615155/Prot_000.pdf